CLINICAL TRIAL: NCT04164134
Title: New Strategies to Detect Cancers in Carriers of Mutations in RB1: Blood Tests Based on Tumor-educated Platelets, or Extracellular Vesicles.
Brief Title: New Strategies to Detect Cancers in Carriers of Mutations in RB1
Acronym: NIRBTEST
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: University Hospital, Essen (Other); Institut Curie (Other); Ligue contre le cancer, France (Other)
Responsible Party: Principal Investigator, Armida W. M. Fabius, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: 129; NL8013 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2019-11-07; First posted 2019-11-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Retinoblastoma; Secondary Primary Malignancies After Retinoblastoma
Keywords: Retinoblastoma; blood test; liquid biopsy; RB1; cancer; Secondary primary malignancies; SPM
MeSH Terms: conditions — Retinoblastoma; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, white blood cells, platelets, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Retinoblastoma patients (children): Children that are currently diagnosed with a retinoblastoma. Blood will be collected and a short questionnaire has to be filled by the parent or legal guardian. Samples will be taken together with standard care blood draw, so no extra venepuncture is required.
  Interventions: Other: blood draw
- Controls (children): Children with an unrelated problem/condition for which surgery is needed Blood will be collected and a short questionnaire has to be filled by the parent or legal guardian. Samples will be taken during standard care blood draw, so no extra venepuncture is required.
  Interventions: Other: blood draw
- Retinoblastoma survivors (adults): Adults that carry a RB1 germline mutation and were diagnosed and treated for retinoblastoma in the past.
  Blood will be collected and a short questionnaire has to be filled.
  Interventions: Other: blood draw
- Controls (adults): Healthy adult controls Blood will be collected and a short questionnaire has to be filled.
  Interventions: Other: blood draw
- Retinoblastoma survivors with Secondary primary malignancies: Adults that carry a RB1 germline mutation, were treated for retinoblastoma in the past, and are currently diagnosed with a secondary primary malignancy.
  Blood will be collected and a short questionnaire has to be filled. Tumor tissue will be collected during surgery.
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — Control samples for the Rb survivor group (adult) are already available at the VUMC for the platelet study; unselected volunteers from an anti-cancer campaign. Control samples (adult) for the EV study will be collected in a blooddrive at the Essen site.
  Pediatric patients. For the pediatric Rb patients, blood draw is part of standard care (3mth-4y). The control blood samples of healthy children (12) will be drawn from healthy children, where the blood draw is already part of otherwise planned care (e.g. patients which are completely healthy besides having an unrelated problem for which surgery is required). Controls will be age-matched as much as possible.

SUMMARY:
Rationale: Individuals with a cancer predisposition due to a mutation in the paradigm tumor suppressor gene RB1, have a high risk to develop the childhood cancer retinoblastoma (Rb). Biopsies are not possible in Rb, before treatment selection. Heritable Rb patients have also a high risk to develop other types of second primary, either childhood or adult, malignancies (SPMs), notably sarcomas and melanomas. Remarkably, SPMs are now the leading cause of death in heritable-Rb-survivors. Unfortunately, there are no well-developed regular surveillance protocols for SPMs in Rb survivors available right now. Recently, new non-invasive cancer test have been developed, based on either RNA-sequencing data from platelets (ThromboSeq), or on extracellular membrane vesicles (EVs) derived from tumor cells present in blood.

Objective:

* Determine the non-cancerous baseline in adult RB1-mutation carriers (heritable-Rb-survivors).
* Contribute to the biobanking of blood and cancerous tissues from RB1-mutation carriers with SPMs.
* The development of blood-based tests, either platelet or EV-based, for the detection of (the type of) tumors in RB1-mutation carriers.

Study design: Cross-sectional multicenter trial.

Study population:

* 40 Rb patients (children),
* 40 controls (children),
* 153 Rb survivors (adults),
* 153 controls (adults),
* 10 Rb survivors with SPM (children/adults).

Main study parameters/endpoints:

* Determine the non-cancerous baseline in adult RB1-mutation carriers (heritable-Rb-survivors).
* Contribute to the biobanking of blood and cancerous tissues from RB1-mutation carriers with SPMs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Two blood samples totalling 10ml blood will be collected for every participant. Additionally, a short questionnaire has to be filled in concerning their and their family's cancer history. Blood draws will be done, when participants are already present in the hospital for other appointments, and thus no extra visits are required. For all children, blood will be collected through an already present IV, and so no extra venepuncture is required. Children have to be included because Rb is a tumor only present in this patient group.

ELIGIBILITY:
Inclusion Criteria:

Adult (16 years and older):

* Group 1: germline mutation RB1.
* Group 2 (control): no germline mutation RB1.

Pediatric (until 6 years of age):

* Group 1: somatic or germline mutation RB1 and retinoblastoma.
* Group 2 (control): no mutation RB1.

Exclusion Criteria:

Adult (16 years and older):

* Group 1: concomitant heritable (inherited) disorder other than caused by monoallelic mutation of RB1.
* Group 2 (control): cancer or already known cancer predisposition syndrome.

Pediatric (until 6 years of age):

* Group 1: concomitant heritable (inherited) disorder other than caused by monoallelic mutation of RB1.
* Group 2: cancer or already known cancer predisposition syndrome.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Control samples for the Rb survivor group (adult) are already available at the VUMC for the platelet study; unselected volunteers from an anti-cancer campaign. Control samples (adult) for the EV study will be collected in a blooddrive at the Essen site.
  Pediatric patients. For the pediatric Rb patients, blood draw is part of standard care (3mth-4y). The control blood samples of healthy children (12) will be drawn from healthy children, where the blood draw is already part of otherwise planned care (e.g. patients which are completely healthy besides having an unrelated problem for which surgery is required). Controls will be age-matched as much as possible.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
RNA expression on platelets and allelic DNA balance of EVs in the blood of adult RB1 mutation carriers (Rb-survivors) and retinoblastoma patients (children). | blood will be taken at study inclusion, patients will be followed throughout the study, max 3 years and 9 months.
  blood analyses at time of inclusion to determine baseline

SECONDARY OUTCOMES:
RNA expression on platelets, allelic DNA balance of EVs in blood and genomic analysis on tumor tissue of RB1-mutation carriers diagnosed with a second primary malignancy. | blood will be taken at study inclusion, patients will be followed throughout the study, max 3 years and 9 months. In case of second primary tumor a second sample will be taken.
  Comparison of blood at time of inclusion and blood at time of SPM diagnosis versus tumor tissue (if available)

CONTACTS AND LOCATIONS:
Overall Officials: Armida Fabius, Principal Investigator — VUMC
Locations (3):
- Institute Curie, Paris, France
- University Hospital Essen (UHE), Essen, Germany
- Amsterdam UMC, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided